CLINICAL TRIAL: NCT02730260
Title: Worksite Phone Counseling for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-1335
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-10

CONDITIONS: Smoking Cessation
Keywords: Directive coaching; Nondirective coaching; smoking cessation quitline; social support
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Directive (Active Comparator): Participants receive up to 7 directive smoking cessation coaching telephone calls from the quitline over 9 weeks.
  Interventions: Behavioral: Directive smoking cessation coaching
- Nondirective (Experimental): Participants receive up to 7 nondirective smoking cessation coaching telephone calls from the quitline over 9 weeks.
  Interventions: Behavioral: Nondirective smoking cessation coaching

INTERVENTIONS:
Behavioral: Nondirective smoking cessation coaching — Quitline coach allows participant to set agenda for each call.
  Arms: Nondirective
Behavioral: Directive smoking cessation coaching — Quitline coach follows a pre-specified agenda for each call, and does not allow participant to deviate from the agenda.
  Arms: Directive

SUMMARY:
Social support is poorly understood but likely to influence outcomes of behavior change efforts. Social support may take a directive or nondirective approach. In directive support, the person attempting a behavior change is told what to do and even what to think. In nondirective support, the person attempting the behavior change decides what to discuss. In some contexts, interactions of race or income with social support have been reported. This is a randomized controlled trial of directive and nondirective coaching in the context of a smoking quitline offered to employees of two large corporations.

DETAILED DESCRIPTION:
BACKGROUND Given the association of smoking with low socioeconomic status, the potential of telephone counseling for smoking cessation to reach diverse audiences needs evaluation. In addition, different approaches to counseling have not been systematically examined, and may differentially affect reach, retention, and success.

PURPOSE To describe employee participation and outcomes in a trial of two counseling styles for telephone-based smoking cessation support.

APPROACH Employees and spouses of two large organizations are invited to participate in a trial of a telephone quitline. Participants are randomized to one of two coaching styles. A protocol-driven (Directive) coaching approach follows a script for each of seven calls over 9 weeks. A participant-centered (Nondirective) coaching approach allowed smokers to select topics of interest, with prompting by the coach as needed. A computer assisted telephone interview program and database provide topics in correct sequence for directive coaching, allow coaches to indicate topics during nondirective coaching, and track time spent on topics in both conditions.

PREDICTOR VARIABLES Demographics, smoking history and conventional self-reported measures of nicotine dependence, smoking urges, preference for patient-centric care, and depression are collected at baseline.

OUTCOMES The primary outcome measure is self-reported abstinence from smoking for 7 days at the time of last follow up, 6 or 12 months after baseline assessment.

ANALYSES Interactions of Race and Income with coaching approach are analyzed. Based on results with asthma patients, a positive interaction of low income with nondirective coaching is tested.

ELIGIBILITY:
Inclusion Criteria:

* Smoking employee or spouse in contemplation, action, or recently entering maintenance stage of change
* English speaking

Exclusion Criteria:

* Smoker in precontemplation stage of change

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2005-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walton Sumner, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers interested in using individual participant data may contact the PI. Only de-identified baseline, 6 month, and 12 month data will be available.

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Sumner W 2nd, Walker MS, Highstein GR, Fischer I, Yan Y, McQueen A, Fisher EB. A randomized controlled trial of directive and nondirective smoking cessation coaching through an employee quitline. BMC Public Health. 2016 Jul 11;16:550. doi: 10.1186/s12889-016-3202-y. PMID 27400966

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 978 persons inquired about the program. 847 took steps to qualify for an employer health insurance discount Of these, 294 declined to enroll, e.g. for being in the precontemplative stage of change.
  553 persons participated in coaching. Of these, 35 worked with coaches in training. 518 participants enrolled in the randomized trial.
Period: Overall Study
Arm/Group | Directive | Nondirective
Started | 258 | 260
Completed | 176 | 185
Not Completed | 82 | 75

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Directive | Nondirective | Total
Number analyzed (Participants) | 258 | 260 | 518
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 252 | 254 | 506
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.3) | 46.0 (10.6) | 46.2 (10.9)
Gender [Count of Participants; unit: Participants]
  Female | 172 | 172 | 344
  Male | 86 | 88 | 174
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 250 | 252 | 502
  Unknown or Not Reported | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 50 | 51 | 101
  White | 199 | 199 | 398
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 258 | 260 | 518
Income [Median (Inter-Quartile Range); unit: units on a scale] — Income levels are:
  1. $0-$15,000
  2. >$15,000-$30,000
  3. >$30,000-$45,000
  4. >$45,000-$60,000
  5. >$60,000-$75,000
  6. >$75,000-$90,000
  7. >$90,000
  units on a scale | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
Education [Median (Inter-Quartile Range); unit: units on a scale] — The education scale is:
  1. Less than 9th grade
  2. 9th grade
  3. 10th grade
  4. 11th grade
  5. High school graduate or General Educational Development (GED)
  6. Some college or trade school
  7. Bachelor's degree
  8. Master's degree
  9. Doctoral degree
  units on a scale | 6 [5 to 7] | 6 [5 to 7] | 6 [5 to 7]
Fagerström Test for Nicotine Dependence (FTND) [Median (Inter-Quartile Range); unit: units on a scale] — Scores for 3 binary and 3 multiple choice items in the Fagerstrom Test for Nicotine Dependence are summed to yield a total score of 0-10.
  .
  Classification of dependence:
  0-2 Very low; 3-4 Low; 5 Moderate; 6-7 High; 8-10 Very high.
  units on a scale | 3 [1 to 5] | 3 [1 to 4] | 3 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence for 7 Days at Last Contact
Description: By self report, the participant has smoked no cigarettes in the past 7 days on the date of last post-intervention assessment, which occurs 6 to 12 months after enrollment.
Time Frame: 6-12 months
Population: These are participants who were successfully contacted at 6 or 12 months following enrollment. Other participants are counted as continuing smokers.
Measure: Number; unit: participants
Arm/Group | Directive | Nondirective
Number analyzed (Participants) | 176 | 185
participants | 68 | 77
Statistical Analysis 1: Comparison: Directive vs Nondirective; Test of the null hypothesis that directive and nondirective coaching have equal smoking cessation rates; Test type: Superiority or Other; p = 0.41, Chi-squared
Statistical Analysis 2: Comparison: Directive vs Nondirective; Odds ratio based on the parameter estimate for the variable, IncomeAboveMedian (0=false, 1=true), from the logistic regression model representing the a priori hypothesis, which specified income, race, and intervention as independent and interacting variables, and smoking cessation at last contact as the dependent variable. An unbalanced variable, PriorQuit (0-=none in the past year, 1=at least one in the past year) was added to the a priori model; Test type: Superiority or Other; p < 0.03, Regression, Logistic; Odds Ratio (OR) = 1.8
Statistical Analysis 3: Comparison: Directive vs Nondirective; Odds ratio for PriorQuit, from the logistic regression model representing the a priori hypothesis, which specified income, race, and intervention as independent and interacting variables, and smoking cessation at last contact as the dependent variable. This variable, PriorQuit (0-=none in the past year, 1=at least one in the past year) was added to the a priori model because it was not balanced after randomization; Test type: Superiority or Other; p < 0.03, Regression, Logistic; Odds Ratio (OR) = 1.6

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Arm/Group | Directive | Nondirective
Serious Adverse Events (participants affected / at risk) | 0/258 | 0/260
Other Adverse Events (participants affected / at risk) | 0/258 | 0/260

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No